CLINICAL TRIAL: NCT00920790
Title: Phase II Clinical Study of KW-0761 in Patients With CCR4-Positive Adult T-cell Leukemia-Lymphoma
Brief Title: Phase II Study of KW-0761 in Subjects With CCR4-positive Adult T-cell Leukemia-lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0761-002
Record Dates: First submitted 2009-06-09; First posted 2009-06-15 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Adult T-cell Leukemia-lymphoma
MeSH Terms: conditions — Leukemia-Lymphoma, Adult T-Cell | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KW-0761 (Experimental)
  Interventions: Biological: KW-0761

INTERVENTIONS:
Biological: KW-0761 — KW-0761 is administered weekly for 8 weeks as an intravenous infusion of 2 hours at a dose of 1.0 mg/kg.
  Other Names: Mogamulizumab

SUMMARY:
To evaluate the efficacy, safety and pharmacokinetic profiles of KW-0761, the anti-CC chemokine receptor 4 (CCR4) antibody, when administered weekly for 8 weeks as an intravenous infusion at a dose of 1.0 mg/kg in relapsed subjects with CCR4-positive adult T-cell leukemia-lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for serum anti-HTLV-I antibody
2. Acute-, lymphoma-, or chronic-type with poor prognostic factors specified in the past
3. Positive for CCR4
4. Relapsed subject after the response (CR, CRu or PR) in the last previous chemotherapy
5. Received at least one prior chemotherapy
6. Subjects with an interval of four weeks or more between the last day of the previous treatment and the scheduled day of the first KW-0761 treatment
7. PS of 0 to 2
8. Negative for HBs antigen and for HBV-DNA by a real-time PCR

Exclusion Criteria:

1. A history of transplantation such as hematopoietic stem cells
2. Positive for HCV antibody or HIV antibody
3. Active multiple cancers at the time of starting this clinical study
4. Previous history of allergic reactions after receiving antibody products
5. Requiring continuous systemic treatment with a steroid
6. Requiring such radiotherapy after starting this clinical study
7. Treated with any investigational drug other than KW-0761 within three months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Result] Ishida T, Joh T, Uike N, Yamamoto K, Utsunomiya A, Yoshida S, Saburi Y, Miyamoto T, Takemoto S, Suzushima H, Tsukasaki K, Nosaka K, Fujiwara H, Ishitsuka K, Inagaki H, Ogura M, Akinaga S, Tomonaga M, Tobinai K, Ueda R. Defucosylated anti-CCR4 monoclonal antibody (KW-0761) for relapsed adult T-cell leukemia-lymphoma: a multicenter phase II study. J Clin Oncol. 2012 Mar 10;30(8):837-42. doi: 10.1200/JCO.2011.37.3472. Epub 2012 Feb 6. PMID 22312108

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 1 June 2009 through 9 November 2010
Groups:
- KW-0761: IV infusions of KW-0761 once/week for 8 weeks at a dose of 1.0mg/kg
Period: Overall Study
Arm/Group | KW-0761
Started | 27
Completed | 13
Not Completed | 14
Not completed — aggravation of general condition | 14

BASELINE CHARACTERISTICS:
Arm/Group | KW-0761
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 64 (7.5) [49 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Response rate defined as the proportion of responders relative to the total population and its exact 95% confidence interval were calculated for best overall response.
  The antitumor response criteria (Complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD)) were created based on the criteria for non-Hodgkin's lymphoma and chronic lymphocytic leukemia provided in the National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology as well as the criteria for non-Hodgkin's lymphoma by the Lymphoma Study Group of the Japan Clinical Oncology Group (JCOG-LSG).Overall Response (OR)= CR + PR.
Time Frame: From date of first subject's consent to participate in the study until the date of last protocol-specified examination for last subject completed, assessed up to 14 months.
Population: Of the 27 subjects enrolled, 26 were included in the efficacy analysis set, whereas 1 was excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | KW-0761
Number analyzed (Participants) | 26
percentage of participants with response | 50 [29.9 to 70.1]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The time from the date of first KW-0761 dosing to the date of progressive disease(PD) confirmation or death.
  The antitumor response criteria including PD were created based on the criteria for non-Hodgkin's lymphoma and chronic lymphocytic leukemia provided in the National Comprehensive Cancer Network(NCCN) Clinical Practice Guidelines in Oncology as well as the criteria for non-Hodgkin's lymphoma by the Lymphoma Study Group of the Japan Clinical Oncology Group (JCOG-LSG).
Time Frame: Baseline to response
Population: Of the 27 subjects enrolled, 26 were included in the efficacy analysis set, whereas 1 was excluded.
Measure: Median (Full Range); unit: days
Arm/Group | KW-0761
Number analyzed (Participants) | 26
days | 97 [12 to 401]

3. Secondary Outcome: Overall Survival (OS)
Description: The time from the date of first KW-0761 dosing to the date of death.
Time Frame: Baseline to response
Population: Of the 27 subjects enrolled, 26 were included in the overall survival analysis set, whereas 1 was excluded.
Measure: Median (Full Range); unit: days
Arm/Group | KW-0761
Number analyzed (Participants) | 26
days | 176.5 [101 to 401]

4. Primary Outcome: Pharmacokinetics-Plasma KW-0761 Concentrations
Description: Statistics of plasma KW-0761 concentrations were tabulated. Individual and mean (+standard deviation) plasma KW-0761 concentrations were plotted on a linear and a logarithmic scale against the time of blood sampling.
  The baseline and maximum time point at which Cmax and Ctrough were collected are 0 to 7 days post-dose.
Time Frame: 0 to 7 days post final dose
Population: Of the 27 subjects enrolled, 27 were included in the pharmacokinetics analysis set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | KW-0761
Number analyzed (Participants) | 27
ng/mL
  Cmax | 42943.2 (14239.5)
  Ctrough | 33638.3 (10572.2)

5. Primary Outcome: Pharmacokinetics-Plasma KW-0761 Concentrations (AUC0-7days)
Description: Statistics of plasma KW-0761 concentrations were tabulated. Individual and mean (+standard deviation) plasma KW-0761 concentrations were plotted on a linear and a logarithmic scale against the time of blood sampling.
Time Frame: 0 to 7 days post final dose
Population: Of the 27 subjects enrolled, 27 were included in the pharmacokinetics analysis set.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | KW-0761
Number analyzed (Participants) | 27
ng·h/mL | 6297408 (1812467)

6. Primary Outcome: Pharmacokinetics-Plasma KW-0761 Concentrations (t1/2)
Time Frame: 0 to 28 days post final dose and follow-up examinations (1 month and 3 months after the end of the post-dosing observation period).
Population: Of the 27 subjects enrolled, 27 were included in the pharmacokinetics analysis set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | KW-0761
Number analyzed (Participants) | 27
hours | 422 (147)

ADVERSE EVENTS:
Arm/Group | KW-0761
Serious Adverse Events (participants affected / at risk) | 6/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KW-0761 (N=27)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Pharyngitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KW-0761 (N=27)
Tachycardia (Cardiac disorders) | 8
Ventricular extrasystoles (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Left atrial dilatation (Cardiac disorders) | 1
Conjunctivitis (Eye disorders) | 1 — Conjunctivitis
Eye pruritus (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 23
Chills (General disorders) | 16
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 2
Application site erythema (General disorders) | 1
Hypothermia (General disorders) | 1
Pain (General disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Nasopharyngitis (Infections and infestations) | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Lymphocyte count decreased (Investigations) | 26
White blood cell count decreased (Investigations) | 18
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 14
Alanine aminotransferase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 11
Blood lactate dehydrogenase increased (Investigations) | 10
Haemoglobin decreased (Investigations) | 8
Blood alkaline phosphatase increased (Investigations) | 7
Blood creatinine increased (Investigations) | 6
Blood pressure increased (Investigations) | 6
Weight increased (Investigations) | 6
Blood albumin decreased (Investigations) | 5
Blood sodium decreased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 4
Weight decreased (Investigations) | 4
Blood pressure decreased (Investigations) | 3
Protein total decreased (Investigations) | 3
Red blood cell count decreased (Investigations) | 3
Blood phosphorus decreased (Investigations) | 3
Blood chloride increased (Investigations) | 2 (2)
Haematocrit decreased (Investigations) | 2 (2)
Blood urine present (Investigations) | 2 (2)
Eosinophil percentage increased (Investigations) | 2 (2)
Blood calcium decreased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Glucose urine present (Investigations) | 1 (1)
Heart rate increased (Investigations) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Mononeuritis (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Disorientation (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Proteinuria (Renal and urinary disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Hot flush (Vascular disorders) | 2
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral circulatory failure (Vascular disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Infusion related reaction (General disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other